CLINICAL TRIAL: NCT02577406
Title: A Phase 3, Multicenter, Open-label, Randomized Study Comparing the Efficacy and Safety of AG-221 (CC-90007) Versus Conventional Care Regimens in Older Subjects With Late Stage Acute Myeloid Leukemia Harboring an Isocitrate Dehydrogenase 2 Mutation
Brief Title: An Efficacy and Safety Study of AG-221 (CC-90007) Versus Conventional Care Regimens in Older Subjects With Late Stage Acute Myeloid Leukemia Harboring an Isocitrate Dehydrogenase 2 Mutation
Acronym: IDHENTIFY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG-221-AML-004
Expanded Access: NCT03723057 (No longer available)
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Results first posted 2022-09-10 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Myeloid; Isocitrate Dehydrogenase
Keywords: AG-221; CC-90007; Efficacy; Safety; Leukemia; Acute myeloid meukemia; Isocitrate dehydrogenase 2 mutation; Enasidenib
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia | interventions — enasidenib; Azacitidine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AG-221 plus Best supportive care (BSC) (Experimental): Continuous 28-day cycles of AG 221 100 mg orally (PO) once a day (QD) for 28 days, plus BSC.
  Interventions: Drug: AG-221; Other: BSC
- Conventional care regimen (CCR) (Active Comparator): Continuous 28-day cycles of BSC only, azacitidine subcutaneously (SC) plus BSC, low-dose cytarabine (LDAC) SC plus BSC, or intermediate-dose cytarabine (IDAC) intravenously (IV) plus BSC. Subjects will be assigned by the investigator to one of the CCR treatment options based on the investigator's assessment of subjects' eligibility.
  Interventions: Other: BSC; Drug: Azacitidine; Drug: Low-dose cytarabine (LDAC); Drug: Intermediate-dose cytarabine (IDAC)

INTERVENTIONS:
Drug: AG-221 — Continuous 28-day cycles of AG 221 100 mg orally (PO) once a day (QD) for 28 days
  Arms: AG-221 plus Best supportive care (BSC)
Other: BSC — Best supportive care includes, hydroxyurea for leukocytosis and/or differentiation-like syndrome, anti-infectives, analgesics, antiemetics, antipyretics, transfusions and nutritional support
Drug: Azacitidine — continuous 28-day cycles of azacitidine 75 mg/m2/day SC for 7 days, plus BSC
  Arms: Conventional care regimen (CCR)
Drug: Low-dose cytarabine (LDAC) — continuous 28-day cycles of cytarabine 20 mg SC twice a day (BID) for 10 days, plus BSC
  Arms: Conventional care regimen (CCR)
Drug: Intermediate-dose cytarabine (IDAC) — 28-day cycles of cytarabine 0.5 to 1.5 g/m2/day IV for 3 to 6 days, per standard institutional practice, plus BSC; only BSC given after IDAC therapy concludes per standard institutional practice
  Arms: Conventional care regimen (CCR)

SUMMARY:
This is an international, multicenter, open-label, randomized, Phase 3 study comparing the efficacy and safety of AG-221 versus conventional care regimens (CCRs) in subjects 60 years or older with acute myeloid leukemia (AML) refractory to or relapsed after second- or third-line AML therapy and positive for an isocitrate dehydrogenase (IDH2) mutation.

DETAILED DESCRIPTION:
Acute myeloid leukaemia (AML) is a form of cancer that is common in older patients. Mutations in the isocitrate dehydrogenase enzyme 2 (IDH2) have been found in approximately 15% of patients with AML.

The outcome of first line chemotherapy treatment is poor and many patients fail to attain complete remission (CR, ie refractory) or will eventually relapse. There is no single standard of care for relapsed or refractory AML. Since the prognosis is very poor there is a great need for new therapies.

Inhibition of the mutant IDH2 enzyme may represent a promising targeted therapy for AML. AG-221 is a small molecule inhibitor of the IDH2 enzyme, designed to preferentially target the mutant IDH2 variants. Data from the ongoing first-in-human study has shown AG-221 to be generally well tolerated and demonstrated CR in patients with IDH2 mutation positive relapsed or refractory AML.

The study purpose is to test the safety and efficacy of AG-221 compared with conventional care regimens (CCR), which include best supportive care (BSC) only, azacitidine plus BSC, low-dose cytarabine plus BSC or intermediate-dose cytarabine plus BSC, in patients with late stage AML refractory to or relapsed after second or third line therapy and positive for the IDH2 mutation. Patients will be randomly assigned to receive open-label tablets of AG-221 or one of the CCR on continuous 28-day treatment cycles. The trial duration is expected to be 78 months which includes 42 months enrollment, approximately 7 months treatment and a follow-up period.

Study procedures include: vital signs, physical exams, ECGs, ECHO, urine/blood samples, bone marrow aspirates and/or biopsies and peripheral blood to test for IDH2 and assess treatment response. Bone marrow, blood, cheek swab samples will be used for genetic tests.

This study is being sponsored by Celgene Corporation. Approximately 316 participants will take part in the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 60 years of age at the time of signing the ICF
2. Subject has primary (ie, de novo) or secondary (progression of MDS or myeloproliferative neoplasms ([MPN], or therapy-related) AML according to WHO classification (Appendix B)
3. Subject has received second- or third-line of AML therapy (see Appendix G for the definition of prior AML line; note that, for subjects having AML secondary to prior higher risk [Intermediate-2 or High risk according to the International Prognostic Scoring System] MDS treated with a hypomethylating agent [eg, azacitidine or decitabine], the hypomethylating therapy can be counted as a line if there is disease progression to AML during or shortly [eg, within 60 days] after the hypomethylating therapy.)
4. Subject has the following disease status:

   1. Refractory to or relapsed after second- or third-line of intensive therapy for AML (eg, the "7 + 3" regimen):

      at least 5% leukemic blasts in bone marrow (the minimum number of treatment cycles of the intensive therapy is per the investigator's discretion); or
   2. Refractory to or relapsed after second- or third-line low-intensity AML therapy (eg, LDAC, azacitidine or decitabine):

   at least 5% leukemic blasts in bone marrow after at least 2 treatment cycles
5. Subject is eligible for and willing to receive the pre-selected CCR treatment option, according to the investigator's assessment (Note: Subjects with degenerative and toxic encephalopathies, especially after the use of methotrexate or treatment with ionizing radiation, should not receive cytarabine.)
6. Subject has Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 (Appendix D)
7. Subject has IDH2 gene mutations tested centrally (using the "investigational use only"PCR assay, Abbott RealTime IDH2) in samples of bone marrow aspirate and peripheral blood, and confirmed positive in bone marrow aspirate and/or peripheral blood. (Note: in the event that the central laboratory result is delayed and precludes acute clinical management of a subject who has confirmed IDH2 gene mutation by local evaluation, the subject may be eligible for randomization with approval by the Medical Monitor.)
8. Subject has adequate organ function defined as:

   * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 3 x upper limit of normal (ULN), unless considered due to leukemic organ involvement, following review by the Medical Monitor; and
   * Serum total bilirubin ≤ 1.5 x ULN, unless considered due to Gilbert's syndrome (eg, a gene mutation in UGT1A1) or leukemic organ involvement, following review by the Medical Monitor; and
   * Creatinine clearance > 30 mL/min based on the Modification of Diet in Renal Disease (MDRD) glomerular filtration rate (GFR):

   GFR (mL/min/1.73 m2) = 175 × (serum creatinine)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American)
9. Females of childbearing potential (FCBP)* may participate, providing they meet the following conditions:

   * Agree to practice true abstinence from sexual intercourse or to use highly effective contraceptive methods (eg, combined [containing estrogen and progestogen] or progestogen-only associated with inhibition of ovulation, oral, injectable, intravaginal, patch, or implantable hormonal contraceptive; bilateral tubal occlusion; intra-uterine device; intrauterine hormone-releasing system; or male partner sterilization [note that vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the FCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success]) at screening and throughout the study, and for 4 months following the last study treatment (6 months following the last dose of cytarabine); and
   * Have a negative serum β-subunit of human chorionic gonadotropin (β-hCG) pregnancy test (sensitivity of at least 25 mIU/mL) at screening; and
   * Have a negative serum or urine (investigator's discretion under local regulations) β-hCG pregnancy test (sensitivity of at least 25 mIU/mL) within 72 hours prior to the start of study treatment in the Treatment Phase (note that the screening serum pregnancy test can be used as the test prior to the start of study treatment in the Treatment Phase if it is performed within the 72-hour timeframe).
10. Male subjects must agree to practice true abstinence from sexual intercourse or to the use of highly effective contraceptive methods (as described above) with non-pregnant female partners of childbearing potential at screening and throughout the course of the study, and should avoid conception with their partners during the course of the study and for 4 months following the last study treatment (6 months following the last dose of cytarabine; 6 months following the last dose of azacitidine in Canada)
11. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted
12. Subject is willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject is suspected or proven to have acute promyelocytic leukemia based on morphology, immunophenotype, molecular assay, or karyotype
2. Subject has AML secondary to chronic myelogenous leukemia
3. Subject has received a targeted agent against an IDH2 mutation
4. Subject has received systemic anticancer therapy or radiotherapy < 14 days prior to the start of study treatment. Note that hydroxyurea is allowed prior to the start of study treatment for the control of leukocytosis (however, hydroxyurea should not be given within 72 hours prior to and after administration of azacitidine).
5. Subject has received non-cytotoxic or investigational agents < 14 days or 5 half-lives, whichever is longer, prior to the start of study treatment
6. Subject has undergone HSCT within 60 days prior to the start of study treatment, or on immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD). The use of a stable dose of oral steroid post-HSCT and/or topical steroids for ongoing skin GVHD is permitted.
7. Subject has persistent, clinically significant non-hematologic toxicities from prior therapies
8. Subject has or is suspected of having central nervous system (CNS) leukemia. Evaluation of cerebrospinal fluid is only required if CNS involvement by leukemia is suspected during screening.
9. Subject has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
10. Subject has immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
11. Subject has significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) class III or IV congestive heart failure (Appendix E); acute coronary syndrome (ACS); and/or stroke; or left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within 28 days prior to the start of study treatment
12. Subject has prior history of malignancy, other than MDS, MPN or AML, unless the subject has been free of the disease for ≥ 1 year prior to the start of study treatment.

    However, subjects with the following history/concurrent conditions are allowed:
    * Basal or squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis clinical staging system)
13. Subject is known seropositive or active infection with human immunodeficiency virus (HIV), or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
14. Subject is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
15. Subjects has uncontrolled hypertension (systolic blood pressure [BP] > 180 mmHg or diastolic BP > 100 mmHg)
16. Subject is a pregnant or lactating female
17. Subject has known or suspected to have hypersensitivity to any of the components of study treatment
18. Subject is taking those medications (listed in Section 8.2) that are known to prolong QT interval unless the subject can be transferred to other medications at least 5 half-lives prior to the start of study treatment
19. Subject has QTc interval (ie, Fridericia's correction [QTcF]) ≥ 450 ms or other factors that increase the risk of QT prolongation or arrhythmic events (eg, heart failure, hypokalemia, family history of long QT interval syndrome) at screening
20. Subject is taking the following sensitive CYP substrate medications that have a narrow therapeutic range are excluded from the study unless the subject can be transferred to other medications at least 5 half-lives prior to the start of study treatment: paclitaxel and docetaxel (CYP2C8), phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline, and tizanidine (CYP1A2)
21. Subject is taking the breast cancer resistance protein (BCRP) transporter-sensitive substrate rosuvastatin should be excluded from the study unless the subject can be transferred to other medications at least 5 half-lives prior to the start of study treatment
22. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
23. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
24. Subject has any condition that confounds the ability to interpret data from the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (93):
- United States (12):
  - Local Institution - 121, Miami, Florida
  - University of Florida Health Cancer Center at Orlando Health, Orlando, Florida
  - Local Institution - 111, Chicago, Illinois
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Local Institution - 128, New York, New York
  - Strong Health System, Rochester, New York
  - Montefiore Medical Center Albert Einstein Cancer Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Local Institution - 104, Greenville, South Carolina
  - Baylor Sammons Cancer Center, Dallas, Texas
- Australia (4):
  - Local Institution - 901, Concord, New South Wales
  - Local Institution - 904, Adelaide, South Australia
  - Local Institution - 906, East Melbourne
  - Local Institution - 905, Melbourne
- Local Institution - 803, Linz, Austria
- Local Institution - 811, Yvoir, Belgium
- Brazil (5):
  - Local Institution - 250, Porto Alegre, Rio Grande do Sul
  - Local Institution - 252, Porto Alegre, RS, Rio Grande do Sul
  - Local Institution - 251, Jaú
  - Local Institution - 253, Rio de Janeiro
  - Local Institution - 254, São Paulo
- Canada (4):
  - Local Institution - 202, Edmonton, Alberta
  - Local Institution - 203, Winnipeg, Manitoba
  - Local Institution - 201, Toronto, Ontario
  - Local Institution - 204, Montreal, Quebec
- China (10):
  - Local Institution - 885, Beijing
  - Local Institution - 884, Beijing
  - Local Institution - 892, Beijing
  - Local Institution - 888, Chengdu, Sichuan
  - Local Institution - 882, Fuzhou
  - Local Institution - 881, Guangzhou, Guangdong
  - Local Institution - 883, Hangzhou
  - Local Institution - 887, Shanghai
  - Local Institution - 891, Shanghai
  - Local Institution - 889, Zhengzhou
- Local Institution - 822, Prague, Czechia
- Denmark (4):
  - Local Institution - 834, Aalborg
  - Local Institution - 833, Arhus C
  - Local Institution - 831, Copenhagen
  - Local Institution - 832, Odense
- France (10):
  - Local Institution - 606, Angers
  - Local Institution - 605, Bobigny
  - Local Institution - 602, Lille
  - Local Institution - 612, Marseille
  - Local Institution - 601, Nantes
  - Local Institution - 607, Pessac
  - Local Institution - 611, Pierre-Bénite
  - Local Institution - 609, Toulouse
  - Local Institution - 610, Versailles
  - Local Institution - 604, Villejuif
- Germany (8):
  - Local Institution - 403, Dresden
  - Local Institution - 413, Essen
  - Local Institution - 406, Frankfurt
  - Local Institution - 401, Hanover
  - Local Institution - 412, Leipzig
  - Local Institution - 402, Mainz
  - Local Institution - 409, München
  - Local Institution - 407, Ulm
- Italy (7):
  - Local Institution - 305, Bologna
  - Local Institution - 304, Brescia
  - Local Institution - 302, Florence
  - Local Institution - 301, Naples
  - Local Institution - 306, Palermo
  - Local Institution - 303, Reggio Calabria
  - Local Institution - 307, Roma
- Russia (4):
  - Local Institution - 861, Krasnoyarsk
  - Local Institution - 864, Moscow
  - Local Institution - 863, Moscow
  - Local Institution - 862, Saint Petersburg
- South Korea (2):
  - Local Institution - 953, Hwasun-gun
  - Local Institution - 952, Seoul
- Spain (6):
  - Local Institution - 701, Oviedo, Principality of Asturias
  - Local Institution - 706, Avda, Campanar 21
  - Local Institution - 708, Barcelona
  - Local Institution - 704, Barcelona
  - Local Institution - 709, Salamanca
  - Local Institution - 702, Seville
- Taiwan (3):
  - Local Institution - 942, Taichung, Northern Dist.
  - Local Institution - 940, Taipei, Zhongzheng Dist.
  - Local Institution - 941, Taoyuan District
- Turkey (Türkiye) (5):
  - Local Institution - 873, Ankara
  - Local Institution - 872, Ankara
  - Local Institution - 871, Ankara
  - Local Institution - 874, Denizli
  - Local Institution - 875, Gaziantep
- United Kingdom (6):
  - Local Institution - 503, Nottingham, Nottinghamshire
  - Local Institution - 501, London
  - Local Institution - 507, London
  - Local Institution - 502, Manchester Withington
  - Local Institution - 510, Oxford
  - Local Institution - 509, Sutton (Surrey)

REFERENCES:
- [Derived] Montesinos P, Fathi AT, de Botton S, Stein EM, Zeidan AM, Zhu Y, Prebet T, Vigil CE, Bluemmert I, Yu X, DiNardo CD. Differentiation syndrome associated with treatment with IDH2 inhibitor enasidenib: pooled analysis from clinical trials. Blood Adv. 2024 May 28;8(10):2509-2519. doi: 10.1182/bloodadvances.2023011914. PMID 38507688
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 319 participants were randomized and 298 participants received treatment
Groups:
- AG-221: Participants receive continuous 28-day cycles of AG-221 100 mg orally (PO) once a day (QD) for 28 days, plus best supportive care (BSC).
- Conventional Care Regimens (CCRs): Treatment options include best supportive care (BSC) only, azacitidine subcutaneous (SC) plus BSC, LDAC subcutaneous (SC) plus BSC, or IDAC intravenously (IV) plus BSC.
  BSC only: Participants receive continuous 28-day cycles of best supportive care (BSC). BSC includes, but is not limited to, hydroxyurea for leukocytosis and/or differentiation syndrome associated with therapy of mutant isocitrate dehydrogenase (IDH) inhibition (ie, IDH differentiation syndrome), anti-infectives, analgesics, antiemetics, antipyretics, transfusions and nutritional support.
  AZA+BSC: Participants receive continuous 28-day cycles of azacitidine 775 mg/m2/day SC for 7 days, plus BSC.
  LDAC+BSC: Participants receive continuous 28-day cycles of cytarabine 20 mg SC twice a day (BID) for 10 days, plus BSC.
  IDAC+BSC: Participants receive 28-day cycles of cytarabine 0.5 to 1.5 g/m2/day IV for 3 to 6 days, per standard institutional practice, plus BSC; only BSC given after intermediate-dose cytarabine (IDAC) therapy concludes per standard institutional practice.
Period: Randomized Period
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Started | 158 | 161
Completed (Continuing to treatment period) | 157 | 141
Not Completed | 1 | 20
Not completed — Death | 1 | 0
Not completed — Other reasons | 0 | 20
Period: Treatment Period
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Started | 157 | 141
Completed | 0 | 0
Not Completed | 157 | 141
Not completed — Death | 38 | 23
Not completed — Adverse Event | 17 | 12
Not completed — Progressive Disease | 53 | 37
Not completed — Withdrawal by Subject | 10 | 24
Not completed — Lost to Follow-up | 0 | 1
Not completed — Transition to commercially available treatment | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Disease Relapse | 28 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Other Reasons | 3 | 39
Not completed — Hematopoietic Stem Cell Transplantation | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AG-221 | Conventional Care Regimens (CCRs) | Total
Number analyzed (Participants) | 158 | 161 | 319
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.4 (6.04) | 70.5 (6.17) | 70.9 (6.11)
Age, Customized [Count of Participants; unit: Participants]
  ≥ 60 to < 70 years | 61 | 72 | 133
  ≥ 70 to < 80 years | 80 | 77 | 157
  ≥ 80 years | 17 | 12 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 65 | 132
  Male | 91 | 96 | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 126 | 128 | 254
  Unknown or Not Reported | 28 | 30 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 12 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 115 | 110 | 225
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 33 | 62

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The time between randomization and death from any cause. Participants who drop-out or are alive at the end of trial will have their OS times censored at the time of last contact, as appropriate.
Time Frame: From randomization to death due to any cause (up to approximately 49 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Months | 6.5 [5.5 to 9.5] | 6.2 [4.6 to 7.7]
Statistical Analysis 1: Comparison: AG-221 vs Conventional Care Regimens (CCRs); Test type: Superiority; p = 0.2288, Stratified Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.67 to 1.10] — The hazard ratio was from a Cox proportional hazards model stratified by prior intensive therapy for AML and primary refractory

2. Secondary Outcome: Overall Response Rate
Description: Number of participants with MLFS + CR + CRi + CRp + PR according to modified International Working Group Acute Myeloid Leukemia (IWG AML) response criteria. Complete response (CR) and morphologic leukemia-free state (MLFS) are defined as <5% blasts in a BM aspirate sample with marrow spicules and a count of ≥200 nucleated cells. There should be no blasts with Auer rods and no extramedullary disease. CR must also include: absolute neutrophil count (ANC) ≥1,000/μL, Platelet count ≥100,000/μL, and independent of red cell transfusions for ≥1 week before each response assessment. Complete remission with incomplete neutrophil recovery (CRi) is all criteria of CR except ANC. Complete remission with incomplete platelet recovery (CRp) is all criteria of CR except platelet count. Partial remission (PR) is defined as all hematologic criteria of CR with a >50% decrease in the percentage of BM blasts to 5% to 25%. (<5% considered if Auer rods are present).
Time Frame: From randomization up to study completion (approximately 78 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Groups:
- Conventional Care Regimens (CCRs): Treatment options include best supportive care (BSC) only, azacitidine subcutaneous (SC) plus BSC, LDAC subcutaneous (SC) plus BSC, or IDAC intravenously (IV) plus BSC.
  BSC only: Participants receive continuous 28-day cycles of best supportive care (BSC). BSC includes, but is not limited to, hydroxyurea for leukocytosis and/or differentiation syndrome associated with therapy of mutant isocitrate dehydrogenase (IDH) inhibition (ie, IDH differentiation syndrome), anti-infectives, analgesics, antiemetics, antipyretics, transfusions and nutritional support.
  AZA+BSC: Participants receive continuous 28-day cycles of azacitidine 775 mg/m2/day SC for 7 days, plus BSC.
  LDAC+BSC: Participants receive continuous 28-day cycles of cytarabine 20 mg SC twice a day (BID) for 10 days, plus BSC.
  IDAC+BSC :Participants receive 28-day cycles of cytarabine 0.5 to 1.5 g/m2/day IV for 3 to 6 days, per standard institutional practice, plus BSC; only BSC given after intermediate-dose cytarabine (IDAC) therapy concludes per standard institutional practice.
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Participants | 64 | 16
Statistical Analysis 1: Comparison: AG-221 vs Conventional Care Regimens (CCRs); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — p-value from a Cochran-Mantel-Haenszel test comparing the response rates between the AG-221 group and the combined CCR group with stratification factors of prior intensive therapy for AML and primary refractory status; Odds Ratio (OR) = 6.08, 95% CI 2-sided [3.32 to 11.14] — Odds ratio from logistic regression

3. Secondary Outcome: Event-Free Survival
Description: Time from randomization to documented morphologic relapse after complete remission/complete remission with incomplete neutrophil recovery/complete remission with incomplete platelet recovery (CR/CRi/CRp), progressive disease (PD) or death from any cause, whichever occurs first. Morphologic Relapse after CR/CRi/CRp is defined as either reappearance of ≥ 5% blasts in the BM not attributable to any other cause or the development of extramedullary disease. PD is defined as a > 50% increase of BM blast count percentage from baseline to ≥ 20% for participants with 5 to 70% BM blasts at baseline or a doubling of absolute blast count in peripheral blood from baseline to ≥ 10 x 109/L (10,000/μL) for participants with > 70% BM blasts at baseline or the development of new extramedullary disease.
Time Frame: From randomization up to study completion (approximately 78 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Months | 4.9 [3.7 to 5.9] | 2.6 [1.9 to 4.4]
Statistical Analysis 1: Comparison: AG-221 vs Conventional Care Regimens (CCRs); Test type: Superiority; p = 0.0200, Stratified Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.55 to 0.95] — The hazard ratio is from a Cox proportional hazards model stratified by prior intensive therapy for AML and primary refractory status

4. Secondary Outcome: Duration of Response
Description: Time from first documented MLFS/CR/CRi/CRp/PR to documented morphologic relapse after CR/CRi/CRp/ PD or death due to any cause, whichever occurs first. CR and MLFS are defined as <5% blasts in a BM aspirate sample with marrow spicules + a count of ≥200 nucleated cells with no blasts with Auer rods + no extramedullary disease. CR must also include: ANC ≥ 1,000/μL, Platelet count ≥100,000/μL, + independent of red cell transfusions for ≥1 week before assessment. CRi is all criteria of CR except ANC. CRp is all criteria of CR except platelet count. PR is defined as all hematologic criteria of CR with >50% decrease in BM blasts to 5%-25%. Relapse after CR/CRi/CRp is defined as reappearance of ≥ 5% blasts in the BM not attributable to other cause or development of extramedullary disease. PD is defined as > 50% increase of BM blast count from baseline to ≥ 20% or a doubling of absolute blast count in peripheral blood from baseline to ≥ 10,000/μL or development of new extramedullary disease.
Time Frame: From randomization up to study completion (approximately 78 months)
Population: All participants who achieved CR/CRi/CRp/PR/MLFS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 64 | 16
Months | 7.4 [5.6 to 12.7] | 33.3 [2.5 to NA] — Not Estimable due to only 6 participants acheiving CR/CRi/CRp/PR/MLFS. For KM methodology to produce an ULN, need 50% of participants to acheive CR/CRi/CRp/PR/MLFS.

5. Secondary Outcome: Time to Response
Description: Time from randomization to first documented MLFS/CR/CRi/CRp/PR. Complete remission (CR) and morphologic leukemia-free state (MLFS) are defined as <5% blasts in a BM aspirate sample with marrow spicules and a count of ≥200 nucleated cells. There should be no blasts with Auer rods and no extramedullary disease. CR must also include the following conditions: absolute neutrophil count (ANC) ≥1,000/μL, Platelet count ≥100,000/μL, and independent of red cell transfusions for ≥1 week before each response assessment. Complete remission with incomplete neutrophil recovery (CRi) is all criteria of CR except ANC. Complete remission with incomplete platelet recovery (CRp) is all criteria of CR except platelet count. partial remission (PR) is defined as all hematologic criteria of CR with a >50% decrease in the percentage of BM blasts to 5% to 25%. (<5% considered if Auer rods are present).
Time Frame: From randomization to to first documented MLFS/CR/CRi/CRp/PR (up to approximately 49 months)
Population: All participants who achieved CR/CRi/CRp/PR/MLFS
Measure: Median (Full Range); unit: Days
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 25 | 7
Days | 58.0 [23 to 242] | 56.0 [27 to 63]

6. Secondary Outcome: Treatment Mortality at 30 Days
Description: The number of participant deaths from any cause within 30 days of initiation of study treatment.
Time Frame: From first dose to 30 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Participants | 10 | 13

7. Secondary Outcome: Treatment Mortality at 60 Days
Description: The number of participant deaths from any cause within 60 days of initiation of study treatment.
Time Frame: From first dose to 60 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Participants | 27 | 30

8. Secondary Outcome: One-Year Survival Rate
Description: The proportion of participants alive at 1 year after randomization
Time Frame: From randomization up to 1 year post (approximately 12 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Proportion of participants | 0.379 [0.303 to 0.454] | 0.263 [0.193 to 0.337]

9. Secondary Outcome: Overall Remission Rate
Description: The number of participants with CR + CRi + CRp according to modified International Working Group Acute Myeloid Leukemia (IWG AML) response criteria. Complete remission (CR) is defined as <5% blasts in a BM aspirate sample with marrow spicules and a count of ≥200 nucleated cells. There should be no blasts with Auer rods and no extramedullary disease. CR must also include the following conditions: absolute neutrophil count (ANC) ≥1,000/μL, Platelet count ≥100,000/μL, and independent of red cell transfusions for ≥1 week before each response assessment. Complete remission with incomplete neutrophil recovery (CRi) is all criteria of CR except ANC. Complete remission with incomplete platelet recovery (CRp) is all criteria of CR except platelet count.
Time Frame: From randomization up to approximately 49 months
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Participants | 47 | 10
Statistical Analysis 1: Comparison: AG-221 vs Conventional Care Regimens (CCRs); Test type: Superiority; p < 0.0001, Fisher Exact

10. Secondary Outcome: Complete Remission Rate
Description: The number of participants with morphologic complete remission (CR) according to modified International Working Group Acute Myeloid Leukemia Response Criteria (IWG AML). CR is defined as less than 5% blasts in a BM aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. There should be no blasts with Auer rods and absence of extramedullary disease; plus the following conditions: absolute neutrophil count (ANC) ≥1,000/μL, Platelet count ≥100,000/μL, and independent of red cell transfusions for ≥1 week before each response assessment.
Time Frame: From randomization up to approximately 49 months
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Participants | 37 | 6
Statistical Analysis 1: Comparison: AG-221 vs Conventional Care Regimens (CCRs); Test type: Superiority; p < 0.0001, Fisher Exact

11. Secondary Outcome: Hematologic Improvement Rate
Description: The number of participants with hematologic improvement neutrophil response (HI-N) + hematologic improvement platelet response (HI-P) + hematologic improvement erythroid response (HI-E) according to the International Working Group for Myelodysplastic Syndromes for Hematologic Improvement (IWG MDS HI) criteria. HI-E is defined as a hemoglobin increase by ≥ 1.5 g/dL and a relevant reduction in units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 week compared with the pretreatment transfusion number in the previous 8 week. HI-P is defined as an absolute increase of ≥ 30 X 10^9/L for participants starting with > 20 X and an increase from < 20 X 10^9/L to > 20 X 10^9/L and by at least 100%. HI-N is defined as At least 100% increase and an absolute increase > 0.5 X 10^9/L.
Time Frame: From randomization up to approximately 49 months
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Participants | 67 | 18
Statistical Analysis 1: Comparison: AG-221 vs Conventional Care Regimens (CCRs); Test type: Superiority; p < 0.0001, Fisher Exact

12. Secondary Outcome: The Number of Participants That Underwent Hematopoietic Stem Cell Transplantation (HSCT)
Description: The number of participants that underwent hematopoietic stem cell transplantation during the study.
Time Frame: From randomization up to approximately 49 months
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Participants | 7 | 2

13. Secondary Outcome: Time to Treatment Failure
Description: Time from randomization to discontinuation of study treatment due to any cause
Time Frame: From randomization to discontinuation of study treatment due to any cause (up to approximately 49 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 158 | 161
Months | 4.9 [4.0 to 6.0] | 1.9 [1.4 to 2.5]
Statistical Analysis 1: Comparison: AG-221 vs Conventional Care Regimens (CCRs); Test type: Superiority; p < 0.0001, Stratified Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.41 to 0.67] — The hazard ratio was from a Cox proportional hazards model stratified by prior intensive therapy for AML and primary refractory status

14. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs)
Description: The number of participants experiencing different types of adverse events (AE). An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. A Serious Adverse Event (SAE) is any AE occurring at any dose that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or constitutes an important medical event. All AEs were coded using the MedDRA Version 22.0. Adverse events were analyzed in terms of treatment-emergent AEs (TEAEs). A treatment-related TEAE was defined as a TEAE that was suspected by the investigator to be related to study treatment. The severity was graded by the study personnel based on NCI National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.
Time Frame: From randomization up to study completion (approximately 78 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 157 | 141
Participants
  Treatment-Emergent Adverse Event (TEAE) | 157 | 131
  TEAE Related to Study Drug | 122 | 86
  Grade ≥ 3 TEAE | 148 | 112
  Grade ≥ 3 TEAE Related to Study Drug | 75 | 49
  Serious TEAE | 139 | 92
  Serious TEAE Related to Study Drug | 34 | 30
  TEAE Leading to Discontinuation of Study Drug | 38 | 16
  Treatment-related TEAE Leading to Discontinuation of Study Drug | 5 | 6
  TEAE Leading to Study Drug Dose Reduction Only | 22 | 3
  Treatment-related TEAE Leading to Study Drug Dose Reduction Only | 18 | 3
  TEAE Leading to Study Drug Dose Interruption Only | 85 | 36
  Treatment-related TEAE Leading to Study Drug Dose Interruption Only | 46 | 21
  TEAE Leading to Study Drug Dose Reduction or Dose Interruption | 92 | 37
  Treatment-related TEAE Leading to Study Drug Dose Reduction or Dose Interruption | 56 | 22
  TEAE Leading to Death | 79 | 33
  Treatment-related TEAE Leading to Death | 1 | 5

15. Secondary Outcome: The Percent of Participants Experiencing Clinically Significant Laboratory Abnormalities - Serum Chemistry
Description: The percent of participants with clinically significant serum chemistry laboratory abnormalities. A clinically significant laboratory abnormality is defined as meeting Grade 3 or Grade 4 criteria according to the Common Terminology Criteria for Adverse Events (CTCAE). Grade 3 is defined as severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care. Grade 4 is defined as life-threatening consequences; urgent intervention indicated. The chemistry panel includes sodium, potassium, calcium, magnesium, chloride, phosphorus, CO2, bicarbonate, blood urea nitrogen (BUN), creatinine, glucose, albumin, total protein, alkaline phosphatase (ALP), bilirubin (total and direct), uric acid, lactate dehydrogenase (LDH), AST/SGOT, ALT/SGPT, gamma glutamyl transpeptidase (GGT), amylase and lipase.
Time Frame: From first dose up to approximately 49 months
Population: All treated participants
Measure: Number; unit: Percent of Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 157 | 141
Percent of Participants | 42.7 | 21.3

16. Secondary Outcome: The Percent of Participants Experiencing Clinically Significant Laboratory Abnormalities - Hematology
Description: The percent of participants with clinically significant hematology laboratory abnormalities. A clinically significant laboratory abnormality is defined as meeting Grade 3 or Grade 4 criteria according to the Common Terminology Criteria for Adverse Events (CTCAE). Grade 3 is defined as severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care. Grade 4 is defined as life-threatening consequences; urgent intervention indicated. The hematology panel includes complete blood count (CBC) with differential, including red blood cell (RBC) count, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), white blood cell (WBC) count (with differential), absolute neutrophil count (ANC) and platelet count.
Time Frame: From first dose up to approximately 49 months
Population: All treated participants
Measure: Number; unit: Percent of Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 157 | 141
Percent of Participants | 94.3 | 89.4

17. Secondary Outcome: The Percent of Participants Experiencing Clinically Significant Vital Sign Abnormalities
Description: The percent of participants with clinically significant vital sign abnormalities including weight, temperature, blood pressure, pulse rate, and respiratory rate.
Time Frame: From first dose up to approximately 49 months
Population: All treated participants
Measure: Number; unit: Percent of Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 157 | 141
Percent of Participants | 0 | 0

18. Secondary Outcome: The Percentage of Participants Experiencing Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: The percent of participants with clinically significant ECG abnormalities. 12-lead ECG was assessed by a physician trained in ECG interpretation. Intervals including PR, QRS, QT and RR were collected, as well as heart rate and rhythm.
Time Frame: From first dose up to approximately 49 months
Population: All treated participants with evaluable measurements
Measure: Number; unit: Percentage of Participants
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 147 | 120
Percentage of Participants | 7.6 | 2.1

19. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire (EORTC QLQ-C30)
Description: The change from baseline in the EORTC QLQ-C30 questionnaire. The EORTC QLQ-C30 is composed of 30 items that address general physical symptoms, physical functioning, fatigue and malaise, and social and emotional functioning. Subscale scores are transformed to a 0 to 100 scale, with higher scores on functional scales indicating better function and higher scores on symptom scales indicating worse symptoms. A change of at least 10 points on the standardized domain scores was required for it to be considered meaningful. Results obtained just prior to the start of study treatment on Day 1 of Cycle 1 will serve as the baseline values. If not available, the most recent screening results prior to the start of study treatment on Day 1 of Cycle 1 will be considered the baseline values.
Time Frame: From baseline to cycle 2 day 1 (up to approximately 1 month)
Population: All participants who completed at least 15 of the 30 items at baseline and at least one post-baseline assessment based on EORTC QLQ-C30
Measure: Mean (Standard Deviation); unit: Change from baseline in QLQ-C30 score
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 106 | 62
Change from baseline in QLQ-C30 score
  Global QoL | -4.7 (20.18) | -4.0 (18.46)
  Physical Functioning | -3.1 (17.19) | -6.7 (21.32)
  Role Functioning | -3.8 (27.63) | -7.8 (29.98)
  Cognitive Functioning | -0.6 (16.89) | -5.1 (18.00)
  Emotional Functioning | 0.9 (15.72) | -0.7 (18.44)
  Social Functioning | -0.6 (29.27) | -10.2 (31.56)
  Fatigue | 5.5 (18.73) | 7.5 (25.59)
  Nausea / Vomiting | 9.0 (20.21) | 1.9 (15.12)
  Pain | 6.0 (23.37) | 7.0 (30.11)
  Dyspnea | -1.3 (23.42) | 0.0 (27.66)
  Insomnia | 8.5 (26.85) | 1.1 (33.04)
  Appetite Loss | 10.7 (28.19) | 8.6 (31.33)
  Constipation | 2.8 (24.82) | 1.6 (24.46)
  Diarrhea | 4.1 (24.21) | 1.6 (18.53)
  Financial Difficulties | -0.3 (24.12) | -3.2 (21.52)

20. Secondary Outcome: Change From Baseline in EQ-5D-5L Health Utility Index
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. These health states are converted to a single index value using the crosswalk method to the EQ-5D-3L value set from the United Kingdom (UK). The EQ-5D-3L health utility index based on the UK population weights range from -0.594 to 1.0 with higher scores indicating higher health utility. Baseline results are obtained just prior to the start of study treatment on Day 1 of Cycle 1 and will serve as the baseline values.
Time Frame: From baseline up to cycle 2 day 1 (up to approximately 1 month)
Population: All participants with non-missing score of EQ-5D-5L Health Utility Index (i.e. all five items were completed) at baseline
Measure: Mean (Standard Deviation); unit: Change from baseline in EQ-5D score
Arm/Group | AG-221 | Conventional Care Regimens (CCRs)
Number analyzed (Participants) | 106 | 62
Change from baseline in EQ-5D score | -0.0738 (0.2128) | -0.0598 (0.2500)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Other (Not Including Serious) Adverse Events were collected form from first dose to study completion (approximately 78 months). All-Cause Mortality was assessed from randomization up to study completion (approximately 99 months).
Description: Serious Adverse Events and Other (Not Including Serious) Adverse Events were assessed/monitored for the treated population. All-Cause Mortality was assessed for the randomized population.
Groups:
- BSC Only: continuous 28-day cycles of BSC
- Azacitidine + BSC: continuous 28-day cycles of azacitidine 75 mg/m2/day SC for 7 days, plus BSC
- LDAC + BSC: continuous 28-day cycles of cytarabine 20 mg SC BID for 10 days, plus BSC
- IDAC + BSC: 28-day cycles of cytarabine 0.5 to 1.5 g/m2/day IV for 3 to 6 days, per standard institutional practice, plus BSC; only BSC given after IDAC therapy concludes per standard institutional practice.
Arm/Group | AG-221 | BSC Only | Azacitidine + BSC | LDAC + BSC | IDAC + BSC
All-Cause Mortality (participants affected / at risk) | 144/158 | 20/22 | 56/69 | 34/37 | 25/33
Serious Adverse Events (participants affected / at risk) | 139/157 | 10/22 | 38/58 | 27/33 | 17/28
Other Adverse Events (participants affected / at risk) | 154/157 | 11/22 | 52/58 | 30/33 | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-221 (N=157) | BSC Only (N=22) | Azacitidine + BSC (N=58) | LDAC + BSC (N=33) | IDAC + BSC (N=28)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 7 | 0 | 0 | 1 | 0
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 33 | 5 | 14 | 13 | 7
HAEMORRHAGIC DISORDER (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
HYPERLEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0
LEUKAEMOID REACTION (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1 | 0
LEUKOSTASIS SYNDROME (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 | 0 | 1 | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
BRADYCARDIA (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CARDIAC HYPERTROPHY (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
RETINAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
GINGIVAL HYPERTROPHY (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
MELAENA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
ODYNOPHAGIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ORAL BLOOD BLISTER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
ASTHENIA (General disorders) | 2 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 4 | 0 | 0 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 14 | 1 | 0 | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1 | 0 | 0
MALAISE (General disorders) | 1 | 0 | 0 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 1 | 0 | 0 | 0 | 0
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 3 | 1 | 1 | 0 | 1
ORGAN FAILURE (General disorders) | 0 | 0 | 1 | 0 | 0
PHYSICAL DECONDITIONING (General disorders) | 1 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 15 | 0 | 2 | 3 | 5
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
CHOLELITHIASIS MIGRATION (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
CHRONIC HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
HEPATIC CYTOLYSIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
HEPATOTOXICITY (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 0 | 0 | 1 | 0 | 0
ACARODERMATITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
ACUTE SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
BACTERAEMIA (Infections and infestations) | 4 | 0 | 0 | 1 | 0
BREVIBACTERIUM INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 0 | 2 | 0 | 0
CAMPYLOBACTER INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 1 | 0 | 0
CLOSTRIDIAL SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 4 | 0 | 1 | 0 | 0
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
COVID-19 PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 0 | 1 | 1 | 0
DISSEMINATED MUCORMYCOSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ENTEROCOCCAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 1 | 0
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
EPIGLOTTITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 1 | 0 | 0 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 2 | 1 | 0 | 0 | 0
FURUNCLE (Infections and infestations) | 0 | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 1 | 0 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
GINGIVITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
HEPATIC INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
HEPATOSPLENIC CANDIDIASIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
HERPES SIMPLEX (Infections and infestations) | 0 | 0 | 1 | 0 | 0
INFECTION (Infections and infestations) | 4 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 2 | 0 | 0 | 1 | 0
INJECTION SITE CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
LIVER ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
MENINGITIS LISTERIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 3 | 0 | 0 | 1 | 0
NOCARDIA SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
NOCARDIOSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTITIS EXTERNA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PERIORBITAL CELLULITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0 | 1 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 27 | 2 | 8 | 4 | 3
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA FUNGAL (Infections and infestations) | 5 | 0 | 2 | 0 | 0
PNEUMONIA INFLUENZAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PSEUDOMONAS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 0 | 0 | 0 | 0
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 0
SEPSIS (Infections and infestations) | 17 | 0 | 3 | 2 | 1
SEPTIC SHOCK (Infections and infestations) | 6 | 2 | 1 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
SKIN INFECTION (Infections and infestations) | 1 | 0 | 2 | 0 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0 | 0 | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
STENOTROPHOMONAS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 1
URETHRITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 4 | 1 | 0 | 1 | 0
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ANAPHYLACTIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
FALL (Injury, poisoning and procedural complications) | 5 | 0 | 2 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
BLAST CELL COUNT INCREASED (Investigations) | 1 | 0 | 2 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
EJECTION FRACTION DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 1 | 0 | 0 | 0 | 0
LIVER FUNCTION TEST INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
TRANSAMINASES INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0 | 0
DIABETIC METABOLIC DECOMPENSATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 | 0 | 0 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 0 | 1 | 1
ACUTE MYELOID LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
DIFFERENTIATION SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 0 | 0 | 0 | 0
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
ONCOLOGIC COMPLICATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
ATAXIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
BRAIN OEDEMA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 4 | 0 | 0 | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
DYSARTHRIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 5 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
LUMBOSACRAL RADICULOPATHY (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 4 | 0 | 1 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 4 | 0 | 3 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
OLIGURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
PURPURA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
HAEMORRHAGE (Vascular disorders) | 1 | 0 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 6 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AG-221 (N=157) | BSC Only (N=22) | Azacitidine + BSC (N=58) | LDAC + BSC (N=33) | IDAC + BSC (N=28)
ANAEMIA (Blood and lymphatic system disorders) | 46 | 2 | 7 | 7 | 7
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 14 | 0 | 7 | 2 | 4
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 20 | 2 | 3 | 3 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 13 | 0 | 3 | 1 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 29 | 2 | 14 | 7 | 4
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 48 | 2 | 17 | 5 | 7
TACHYCARDIA (Cardiac disorders) | 2 | 2 | 1 | 1 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 4 | 0 | 1 | 2 | 0
DRY EYE (Eye disorders) | 4 | 0 | 4 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 10 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 17 | 0 | 5 | 2 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 11 | 2 | 4 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 30 | 2 | 23 | 4 | 6
DIARRHOEA (Gastrointestinal disorders) | 62 | 0 | 14 | 7 | 6
DRY MOUTH (Gastrointestinal disorders) | 2 | 0 | 3 | 2 | 0
DYSPEPSIA (Gastrointestinal disorders) | 9 | 1 | 1 | 1 | 1
GINGIVAL BLEEDING (Gastrointestinal disorders) | 11 | 1 | 2 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 5 | 1 | 5 | 1 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 10 | 1 | 3 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 69 | 2 | 16 | 10 | 7
STOMATITIS (Gastrointestinal disorders) | 15 | 1 | 4 | 7 | 5
VOMITING (Gastrointestinal disorders) | 40 | 1 | 9 | 5 | 1
ASTHENIA (General disorders) | 29 | 2 | 13 | 5 | 4
FATIGUE (General disorders) | 45 | 0 | 10 | 6 | 4
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 10 | 1 | 0 | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 5 | 0 | 3 | 0 | 0
INJECTION SITE PAIN (General disorders) | 0 | 0 | 6 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 5 | 1 | 3 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 33 | 1 | 13 | 6 | 2
PYREXIA (General disorders) | 37 | 4 | 14 | 5 | 5
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 15 | 0 | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 3 | 0 | 0 | 2 | 1
CELLULITIS (Infections and infestations) | 3 | 1 | 2 | 2 | 1
INFECTION (Infections and infestations) | 2 | 0 | 1 | 0 | 2
ORAL CANDIDIASIS (Infections and infestations) | 10 | 1 | 2 | 1 | 0
PHARYNGITIS (Infections and infestations) | 3 | 0 | 0 | 2 | 0
PNEUMONIA (Infections and infestations) | 13 | 1 | 7 | 0 | 2
PNEUMONIA FUNGAL (Infections and infestations) | 3 | 0 | 3 | 0 | 0
RHINITIS (Infections and infestations) | 4 | 0 | 3 | 0 | 1
TOOTH INFECTION (Infections and infestations) | 2 | 0 | 0 | 2 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 | 0 | 6 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 12 | 2 | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 12 | 0 | 3 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 13 | 0 | 4 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 | 0 | 3 | 2 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 | 0 | 1 | 1 | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 | 0 | 3 | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 41 | 0 | 1 | 1 | 2
BLOOD CREATININE INCREASED (Investigations) | 20 | 0 | 5 | 0 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 8 | 0 | 4 | 3 | 1
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 8 | 0 | 3 | 0 | 0
WEIGHT DECREASED (Investigations) | 14 | 0 | 4 | 1 | 2
WEIGHT INCREASED (Investigations) | 0 | 0 | 0 | 1 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 49 | 1 | 13 | 5 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 11 | 0 | 1 | 1 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 3 | 0 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 17 | 0 | 1 | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 13 | 2 | 4 | 0 | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 15 | 0 | 3 | 0 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 52 | 1 | 10 | 2 | 7
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 19 | 1 | 3 | 2 | 6
HYPONATRAEMIA (Metabolism and nutrition disorders) | 10 | 0 | 2 | 1 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 9 | 0 | 3 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13 | 1 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 21 | 0 | 3 | 2 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 11 | 1 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 20 | 0 | 6 | 5 | 1
DIFFERENTIATION SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 0 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 23 | 0 | 0 | 1 | 0
DYSGEUSIA (Nervous system disorders) | 12 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 24 | 0 | 3 | 5 | 2
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 4 | 0 | 3 | 1 | 0
ANXIETY (Psychiatric disorders) | 9 | 0 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 9 | 0 | 0 | 2 | 2
DEPRESSION (Psychiatric disorders) | 8 | 0 | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 24 | 1 | 10 | 2 | 2
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 2 | 0 | 3 | 1 | 0
DYSURIA (Renal and urinary disorders) | 2 | 0 | 3 | 0 | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 27 | 3 | 9 | 8 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 34 | 2 | 3 | 3 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 27 | 3 | 10 | 4 | 4
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 2 | 4 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 3 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 6 | 0 | 5 | 1 | 1
PETECHIAE (Skin and subcutaneous tissue disorders) | 13 | 0 | 4 | 4 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 13 | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 11 | 0 | 6 | 0 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 9 | 0 | 1 | 1 | 1
HAEMATOMA (Vascular disorders) | 11 | 0 | 2 | 0 | 0
HYPERTENSION (Vascular disorders) | 8 | 0 | 4 | 1 | 2
HYPOTENSION (Vascular disorders) | 15 | 0 | 1 | 0 | 1
PHLEBITIS (Vascular disorders) | 2 | 1 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT02577406/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT02577406/SAP_001.pdf